CLINICAL TRIAL: NCT06096285
Title: Heterogeneity and Disease Development of Early Chronic Obstructive Pulmonary Disease
Brief Title: Heterogeneity and Development of Early COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jieping LEI, Ph.D., Principal Investigator, China-Japan Friendship Hospital
Other Study IDs: 2023-ZF-9
Record Dates: First submitted 2023-10-15; First posted 2023-10-23 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic obstructive pulmonary disease; Early COPD; Heterogeneity; Disease development
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Preserved ratio impaired spirometry (PRISm): People with post-bronchodilator forced expiratory volume in one second (FEV1)/forced vital capacity (FVC) ≥ 0.70 and FEV1 and/or FVC < 80% predicted, or FEV1/FVC ≥ lower limit of normal (LLN) and FEV1 < LLN.
- COPD Stage 0: People who had COPD-related risk factor exposure (e.g. cigarette smoke) and/or presented with respiratory symptoms (e.g. chronic cough, and/or sputum production) whereas with normal pulmonary function.
- Pre-COPD: People (importantly, of any age) who had respiratory symptoms (e.g. cough, sputum production, dyspnea, and/or exacerbation) with or without detectable structural (e.g. thoracic computed tomography (CT) emphysema, small and/or large airway impairments) and/or functional (e.g. low diffusion capacity for carbon monoxide (DLCO), hyperinflation, small airway obstruction, and/or accelerated FEV1 decline) abnormalities, in the absence of airflow limitation, and who might (or not) develop persistent airflow limitation (i.e. COPD) over time.
- Early COPD: People who were younger than 50 years with ten or more pack-years smoking history and any of these abnormalities: i) early airflow limitation (post-bronchodilator FEV1/FVC < LLN), ii) compatible thoracic CT abnormalities, iii) rapid decline in FEV1 (> 60 ml/year) that was accelerated relative to FVC.
- Young COPD: COPD patients with post-bronchodilator FEV1/FVC < 0.70 diagnosed in the 20-50 year age range.
- Mild COPD: COPD patients with post-bronchodilator FEV1/FVC < 0.70 and FEV1 ≥ 80% predicted.
- Controls: People who were not belonged to any of above six early COPD status, and with pre- and post-bronchodilator FEV1/FVC ≥ 0·70, and with post-bronchodilator FEV1/FVC ≥ LLN.

SUMMARY:
This study aims to investigate the clinical characteristics and heterogeneities of early chronic obstructive pulmonary disease (COPD), to determine the disease development of early COPD, and to establish a multidimensional model for predicting the outcomes of early COPD.

ELIGIBILITY:
Inclusion Criteria:

* The individuals who meet the defining criteria of PRISm, COPD Stage 0, Pre-COPD, Early COPD, Young COPD, and Mild COPD, according to the latest GOLD documents and publications.

Exclusion Criteria:

* Age < 18 years or > 80 years;
* Pregnant or maternal women;
* Having malignant and active tumor(s), and receiving treatment;
* Undergoing a surgical operation;
* Having problems with mental awareness;
* Having difficulties in daily activities;
* Participating in other interventional clinical trials.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study plans to involve the individuals with different early COPD status, as well as comparable controls.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with COPD exacerbation | One year
  COPD exacerbation refers to acute deterioration of respiratory symptoms (e.g. cough, sputum, wheeze, dyspnea), especially resulting in hospital visit or admission.

SECONDARY OUTCOMES:
FEV1 | One year
FVC | One year
FEV1/FVC ratio | One year
FEV1% predicted value | One year
FVC% predicted value | One year
The COPD Assessment Test scale | One year
  The COPD Assessment Test scores range from 0 to 40, with higher scores indicating worse symptoms.
The modified Medical Research Council dyspnea scale | One year
  The modified Medical Research Council dyspnea scores range from 0 to 4, with higher scores indicating more severe dyspnea.

CONTACTS AND LOCATIONS:
Overall Officials: Jieping Lei, Ph.D., Principal Investigator — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No